CLINICAL TRIAL: NCT00037232
Title: Failure Time Methods for Family Disease Studies
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 1140; R01HL065411 (NIH)
Record Dates: First submitted 2002-05-16; First posted 2002-05-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2005-05

CONDITIONS: Heart Diseases; Cardiovascular Diseases; Coronary Disease
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Coronary Disease

SUMMARY:
To develop statistical methodologies to study genetic and environmental factors in cardiovascular disease, using age at onset data from population-based family studies of disease incidence.

DETAILED DESCRIPTION:
BACKGROUND:

In the study of chronic diseases, both environmental and genetic factors can be influential. In highly common diseases, such as coronary heart disease, genetic effects may be more influential in determining the age of onset of the disease than in determining whether or not one gets the disease. When sufficient information is available, family studies can help localize possible disease genes on the human chromosome through genetic linkage analysis, and familial aggregation of disease can help separate the effects of inheritance, environment and lifestyle on the risk of disease.

DESIGN NARRATIVE:

The study developed: (1) a general strategy for evaluating the fit of parametric dependence models for familial clustering of ages at disease-onset; (2) a computationally simple method for genetic linkage analysis of age at onset data; (3) application and illustration of recently developed additive frailty models for complex familial dependence structures. Method (1) was applied to a family study of cardiovascular disease and a twin study of appendectomy. Method (2) was applied to ongoing genetic studies conducted at the University of California at San Francisco. Method (3) was applied to a family study of coronary heart disease in Western Australia. Well-documented, user-friendly programs were developed and made publicly available.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-04; Study Completion 2005-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Glidden — University of California at San Francisco

REFERENCES:
- [Background] Glidden DV. Robust inference for event probabilities with non-Markov event data. Biometrics. 2002 Jun;58(2):361-8. doi: 10.1111/j.0006-341x.2002.00361.x. PMID 12071409
- [Background] St Jeor ST, Perumean-Chaney S, Sigman-Grant M, Williams C, Foreyt J. Family-based interventions for the treatment of childhood obesity. J Am Diet Assoc. 2002 May;102(5):640-4. doi: 10.1016/s0002-8223(02)90146-x. No abstract available. PMID 12008987
- [Background] Glidden DV, Liang KY, Chiu YF, Pulver AE. Multipoint affected sibpair linkage methods for localizing susceptibility genes of complex diseases. Genet Epidemiol. 2003 Feb;24(2):107-17. doi: 10.1002/gepi.10215. PMID 12548672
- [Background] Glidden DV, Liang KY. Ascertainment adjustment in complex diseases. Genet Epidemiol. 2002 Oct;23(3):201-8. doi: 10.1002/gepi.10204. PMID 12384971
- [Background] Glidden DV, Vittinghoff E. Modelling clustered survival data from multicentre clinical trials. Stat Med. 2004 Feb 15;23(3):369-88. doi: 10.1002/sim.1599. PMID 14748034